CLINICAL TRIAL: NCT06992362
Title: Prospective, Single-arm, Single-center Phase II Clinical Study of Perioperative Precision Treatment for Locally Advanced Hepatoid Adenocarcinoma of Stomach
Brief Title: Perioperative Treatment of Hepatoid Adenocarcinoma of Stomach
Acronym: HASCHANGE01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH2024296
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Hepatoid Adenocarcinoma of Stomach
Keywords: HER2; SOX; PD-1 inhibitor; Disitamab Vedotin; perioperative treatment

STUDY DESIGN:
Intervention Model Description: perioperative treatment with Disitamab Vedotin，SOX and Sintilimab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- perioperative treatment for hepatoid adenocarcinoma of stomach (Experimental): 1. Neoadjuvant therapy: Disitamab Vedotin 2.5mg/kg, d1, a course of treatment every 21 days; Sindilizumab 200mg intravenously, d1, every 21 days; Tegafur,Gimeracil and Oteracil Porassium Capsules (by body surface area: BSA<1.25m2, 40mg; BSA≥1.25m2, <1.5m2, 50mg; BSA≥1.5m2,60mg), orally, twice a day, d1-14, every 21 days; Oxaliplatin 85mg/m2, IV, d1, every 21 days.
  2. Radical surgical treatment should be performed within 4-6 weeks after the end of neoadjuvant therapy.
  3. Adjuvant therapy: Adjuvant therapy begins within 4-6 weeks after surgery. Disitamab Vedotin 2.5mg/kg intravenously, d1, one course every 21 days; Sindilizumab 200mg intravenously, d1, every 21 days; Tegafur,Gimeracil and Oteracil Porassium (by body surface area:BSA<1.25m2, 40mg; BSA≥1.25m2, <1.5m2, 50mg; BSA≥1.5m2,60mg) orally, 2 times daily, d1-14, one course every 21 days.
  Interventions: Drug: Perioperative treatment

INTERVENTIONS:
Drug: Perioperative treatment — RC48+SOX+Sindilizumab

SUMMARY:
The goal of this clinical trial is to learn if treatment modality including Disitamab Vedotin （RC48）, Oxaliplatin，Tegafur,Gimeracil and Oteracil Porassium Capsules （SOX）and Sindillimab works to treat locally advanced hepatoid adenocarcinoma of stomach. It will also learn about the safety of this modality. The main aim it aims to achieve are:

* To evaluate the perioperative efficacy of RC48 combined with sindillizumab and SOX in the treatment of locally advanced HER2-expressing hepatoid adenocarcinoma of stomach
* To evaluate the safety and long-term benefits of RC48 combined with sindillizumab and SOX regimens in perioperative treatment of locally advanced HER2-expressing hepatoid adenocarcinoma of stomach

Participants will:

* Preoperative treatment with RC48, SOX and sindillizumab for 4 cycles
* Radical surgery after 4-6 weeks of the preoperative treatment
* Adjuvant treatment with RC48, Tegafur,Gimeracil and Oteracil Porassium Capsules and sindillizumab for 4 cycles

ELIGIBILITY:
Inclusion Criteria:

* The histological type of gastric hepatoid adenocarcinoma was confirmed by pathological biopsy；
* HER2 expression (Immunohistochemistry: 1+,2+,3+);
* Patients with clinical stage II-III;
* Those who are expected to complete R0 excision;
* ECOG score 0~1;
* Generally in good condition, perioperative treatment and surgical resection can be tolerated;
* Patients were enrolled voluntarily.

Exclusion Criteria:

* Combined with other malignant tumors (excluding thyroid papillary carcinoma, facial basal cell carcinoma and other low-grade malignant tumors); -Patients with obstruction, bleeding, etc. who need surgical intervention after evaluation by clinicians;
* dMMR/MSIH status；
* Received other anti-tumor therapy before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | within 10 days after surgery
  The proportion of subjects with node-negative lymph nodes and without residual viable tumor cells in the total number of subjects

SECONDARY OUTCOMES:
major pathological response rate | within 10 days after surgery
  The proportion of subjects with surviving tumor cells ≤10% in total subjects;
Objective response rate | From enrollment to surgery, assessed up to 3 months
  Proportion of patients who achieved pre-defined tumor volume reduction , including patients with complete response (CR) and partial response (PR).
Event-free survival | From date of enrollment until the date of first documented progression, recurrence or date of death from any cause, whichever came first, assessed up to 3 years
  From the start of treatment to the first occurrence of any of the following events: disease progression without surgical treatment, local or distant recurrence, death from any cause
Disease free survival | From date of surgery until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 3 years
  It usually starts from the time when the patient receives treatment (such as surgery), and ends at the time when the disease recurs (such as tumor recurrence, metastasis) or when the patient dies for any reason
overall survival | From date of diagnosis until the date of death from any cause, assessed up to 3 years
  It refers to the period from when the patient is diagnosed until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: jiafu ji, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after the publication of the results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the publication